CLINICAL TRIAL: NCT03852576
Title: Phase 1B In-vivo Study of KSP/QRH Heptapeptide Dimer for Detection of Neoplasia in the Esophagus
Brief Title: Phase 1B Study of KSP/QRH Dimer for Detection of Neoplasia in the Esophagus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study had to be terminated for lack of dimer and inability to produce more at this time.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Danielle Kim Turgeon, Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00158121
Record Dates: First submitted 2019-02-20; First posted 2019-02-25 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Esophagus sprayed with KSP/QRH dimer (Experimental): Area of interest in subject's esophagus sprayed with KSP/QRH dimer and imaged with the SFE probe
  Interventions: Drug: KSP/QRH dimer

INTERVENTIONS:
Drug: KSP/QRH dimer — KSP-QRH-E3-IRDye800 (Peptide 919288G)

SUMMARY:
The overall aim of this feasibility study is to develop new technologies for improved detection of Barrett's neoplasia using the scanning fiber endoscope (SFE) imaging system. This study will combine the use of a fluorescent-labeled peptide dimer that bind specifically to pre-cancerous mucosa in the esophagus for use as a novel imaging agent to guide endoscopic biopsy or endoscopic mucosal resection (EMR). This Phase 1B study will be used to provide early evidence of efficacy for the topical application of a peptide dimer that binds to molecular targets, including EGFR and HER2, that are specific for esophageal dysplasia. A dimer is needed because cancer in the esophagus is genetically heterogeneous. QRH binds specifically to Epidermal Growth Factor Receptor (EGFR), and KSP binds specifically to Human Epithelial Growth Factor Receptor (HER2). The study will look at peptide binding in subjects with known or suspected Barrett's esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Has known or suspected Barrett's esophagus
* Scheduled for a clinically-indicated, upper endoscopy
* Subject is medically cleared for the procedure (e.g. washout for anticoagulants, co-morbidities)
* Age 18 to 100 years
* Willing and able to sign informed consent

Exclusion Criteria:

* Subjects with known allergy or negative reaction to the near infrared fluorophore IRDye800CW, or derivatives
* Subjects on active chemotherapy or radiation treatment
* Pregnant or trying to conceive

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Binding of KSP/QRH dimer to EGFR and HER2 | During and immediately after procedure, generally no more than 2 hours
  Validation of the dimer to EGFR and HER2 using target-to-background ratio of the suspicious region compared to the background
SFE ability to detect dimer by SNR | During and immediately after procedure, generally no more than 2 hours
  SFE (scanning fiber endoscope) imaging system will be used to image the dimer on the area of interest using signal-to-noise ratio (SNR)
SFE ability to detect dimer by fluorescence T/B ratio | During and immediately after procedure, generally no more than 2 hours
  SFE (scanning fiber endoscope) imaging system will be used to image the dimer on the area of interest using fluorescence tumor-to-background (T/B) ratio
SFE ability to detect dimer with contrast | During and immediately after procedure, generally no more than 2 hours
  SFE (scanning fiber endoscope) imaging system will be used to image the dimer on the area of interest using contrast

CONTACTS AND LOCATIONS:
Overall Officials: Danielle K Turgeon, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chen J, Jiang Y, Chang TS, Rubenstein JH, Kwon RS, Wamsteker EJ, Prabhu A, Zhao L, Appelman HD, Owens SR, Beer DG, Turgeon DK, Seibel EJ, Wang TD. Detection of Barrett's neoplasia with a near-infrared fluorescent heterodimeric peptide. Endoscopy. 2022 Dec;54(12):1198-1204. doi: 10.1055/a-1801-2406. Epub 2022 Mar 17. PMID 35299273